CLINICAL TRIAL: NCT03894085
Title: Definitive Selection of Neuroimaging Biomarkers in Anxiety Disorder and Obsessive-compulsive Disorder: A Longitudinal Functional Magnetic Resonance Imaging （ fMRI ）Study With Paroxetine Treatment
Brief Title: Definitive Selection of Neuroimaging Biomarkers in Anxiety Disorder and Obsessive-compulsive Disorder: A Longitudinal Functional Magnetic Resonance Imaging （fMRI） Study With Paroxetine Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Guo Wenbin, Professor of Psychiatry Department of Psychiatry of the Second Xiangya Hospital, Central South University, Central South University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016YFC1307104
Record Dates: First submitted 2019-03-18; First posted 2019-03-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Disorder; Obsessive-Compulsive Disorder
Keywords: anxiety disorder; obsessive-compulsive disorder; neuroimaging; biomarkers; treatment response
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GAD group (Experimental): 1. General anxiety disorder(GAD) patients meet the diagnostic criteria of the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-V)
  2. MRI scan and evaluation of clinical symptoms at baseline and 4 weeks
  3. Paroxetine (20-40mg) treatment for 4 weeks
  Interventions: Drug: Paroxetine
- PD group (Experimental): 1. Panic disorder(PD) patients meet the diagnostic criteria of the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-V)
  2. MRI scan and evaluation of clinical symptoms at baseline and 4 weeks
  3. Paroxetine (20-40mg)treatment for 4 weeks
  Interventions: Drug: Paroxetine
- SAD group (Experimental): 1. Social anxiety disorder(SAD)meet the diagnostic criteria of the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-V)
  2. MRI scan and evaluation of clinical symptoms at baseline and 4 weeks
  3. Paroxetine (20-40mg)treatment for 4 weeks
  Interventions: Drug: Paroxetine
- OCD group (Experimental): 1. Obsessive-compulsive disorder (OCD)meet the diagnostic criteria of the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-V)
  2. MRI scan and evaluation of clinical symptoms at baseline and 4 weeks
  3. Paroxetine(40-80mg) treatment for 4 weeks
  Interventions: Drug: Paroxetine
- Healthy controls (No Intervention): MRI scan at baseline and no drugs treatment

INTERVENTIONS:
Drug: Paroxetine — Paroxetine treatment for 4 weeks usage:20-80mg Qd
  Arms: GAD group; OCD group; PD group; SAD group

SUMMARY:
To explore reliable neuroimaging biomarkers for anxiety disorder and OCD,and whether there are shared imaging biomarkers between different subtypes of anxiety disorder and OCD, the investigators included30 drug-naive general anxiety disorder (GAD),30 drug-naïve panic disorder(PD),30 drug-naïve social anxiety disorder,30 drug-naive.obsessive-compulsive disorder patients and 30 healthy controls by using a combination of cross-section and longitudinal study designs, including a longitudinal study in patients with anxiety disorder and OCD with 4 weeks of selective serotonin reuptake inhibitor (SSRI) paroxetine treatment. The investigators will also evaluate the severity of symptom, social function, cognitive function and treatment response.

DETAILED DESCRIPTION:
Previous studies suggest that there are brain anatomical and functional in patients with anxiety disorder and obsessive-compulsive disorder (OCD). However, it remains unclear whether these abnormalities can be used for the diagnosis of anxiety disorder、OCD and prediction of treatment effects. It is also unclear whether there are shared imaging biomarkers between different subtypes of anxiety disorder and OCD.And it still lacks reliable neuroimaging biomarkers in anxiety disorder and OCD. Based on the previous studies, this study aims to examine the whole-brain anatomical and functional abnormalities in 30 general anxiety disorder (GAD),30 panic disorder(PD),30 social anxiety disorder,30 obsessive-compulsive disorder patients and 30 healthy controls by using a combination of cross-section and longitudinal study designs, including a longitudinal study in patients with anxiety disorder and OCD with 4 weeks of selective serotonin reuptake inhibitor (SSRI) paroxetine treatment.First, neuroimaging biomarkers are definitively selected in subjects at different subtypes of anxiety disorder and OCD population for the purpose of diagnosis by using a cross-section design. After that, a longitudinal study is conducted in patients with anxiety disorder and OCD with 4 weeks of paroxetine treatment to validate that the selected neuroimaging biomarkers can be used to predict treatment response of medication. The definitively selected neuroimaging biomarkers are expected to be useful for the diagnosis of anxiety disorder and OCD, and prediction of treatment effects; and finally be helpful for understanding the pathophysiology of anxiety disorder and OCD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for GAD、PD、SAD、OCD patients according to the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-V)
* Never received any treatment before,and with no psychotic symptoms
* For Healthy controls:Their ﬁrst-degree relatives had no history of psychiatric disorders

Exclusion Criteria:

* Exclusion criteria for all participants were any other psychiatric diagnoses according to DSM-V; any physical illness such as liver and kidney diseases, cardiovascular diseases; any combined with other antipsychotic medications (both low and high doses), including typical and atypical antipsychotic,mood stabilizer, antidepressant drugs ; history of drug or alcohol abuse or dependence; obvious suicide attempts or behaviors; pregnancy or lactation. and any contraindications to MRI scan.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
structural and function MRI data | 4 weeks
  A 3.0 T Siemens scanner was used to obtain the fMRI images in the Second Xiangya Hospital of Central South University.The MRI data wii be obtained before and after treatment at different follow up point.
Hamilton anxiety scale(HAMA) | 4 weeks
  The change of the Hamilton anxiety scale(HAMA) total score, severity of anxiety symptoms before and after treatment at different follow up point.
Yale-Brown Obsessive Compulsive Scale(Y-BOCS) | 4 weeks
  The change of the Yale-Brown Obsessive Compulsive Scale(Y-BOCS)total score, severity of obsessive-compulsive symptom before and after treatment at different follow up point.
Brief Cognitive Assessment Tool for Schizophrenia (B-CATS) | 4 weeks
  The investigators will use the Brief Cognitive Assessment Toolfor Schizophrenia (B-CATS) score as primary assess of cognitive function before and after treatment at different follow up point.

SECONDARY OUTCOMES:
Social Disability Screening Schedule(SDSS) | 4 weeks
  The investigators will use the Social Disability Screening(SDSS) score as assess of social function before and after treatment at different follow up point.
Simplified Coping Style Questionnaire (SCSQ) | 4 weeks
  The investigators will use the Simplified Coping Style Questionnaire(SCSQ) scale score as assess of coping style at baseline and after 4 weeks
Eysenck Personality Questionnaire(EPQ) | at baseline
  The investigators will use the Eysenck Personality Questionnaire (EPQ) scale as assess of characteristic of personality at baseline
The 17-item Hamilton depression scale (HAMD-17) | 4 weeks
  The change of the 17-item Hamilton depression scale total score, severity of depressive symptom before and after treatment at different follow up point
Liebowitz social anxiety scale(LSAS) | 4 weeks
  The change of the Liebowitz social anxiety scale (LSAS) total score,severity of social anxiety before and after treatment at different follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Guo, MD Ph.D, Principal Investigator — Central South University; Xiaoxiao Shan, M.D, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, China

REFERENCES:
- [Derived] Han Y, Yan H, Shan X, Li H, Liu F, Li P, Zhao J, Guo W. Shared and distinctive neural substrates of generalized anxiety disorder with or without depressive symptoms and their roles in prognostic prediction. J Affect Disord. 2024 Mar 1;348:207-217. doi: 10.1016/j.jad.2023.12.067. Epub 2023 Dec 29. PMID 38160885
- [Derived] Han Y, Yan H, Shan X, Li H, Liu F, Li P, Zhao J, Guo W. Disrupted functional connectivity associated with cognitive impairment in generalized anxiety disorder (GAD) and comorbid GAD and depression: a follow-up fMRI study. J Psychiatry Neurosci. 2023 Nov 7;48(6):E439-E451. doi: 10.1503/jpn.230091. Print 2023 Nov-Dec. PMID 37935477